CLINICAL TRIAL: NCT03310476
Title: Influence of Resistant Starch in Baked and Boiled Potatoes on Glycemic and Satiety Responses in Overweight Females
Brief Title: Influence of Resistant Starch Intake in Potatoes on Blood Glucose and Satiety Responses in Overweight Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Principal Investigator, Mindy Patterson Maziarz, Assistant Professor, Texas Woman's University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Resistant starch in potatoes
Record Dates: First submitted 2017-09-21; First posted 2017-10-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baked, consumed chilled potatoes (Experimental)
  Interventions: Other: Potatoes
- Boiled, consumed hot potatoes (Experimental)
  Interventions: Other: Potatoes

INTERVENTIONS:
Other: Potatoes — Participants will follow the same protocol for each arm with a minimum of 1-week wash-out period between arms. For each arm, fasting blood will be collected then 200 g of potato will be consumed. Postprandial blood will be collected 15, 30, 60, and 120 minutes. Subjective satiety will be assessed using Visual Analogue Scale three times, as well as 48-hour subsequent dietary intake.

SUMMARY:
Resistant starch (RS) is a type of fiber that has unique digestive properties that can impact overall health including glucose homeostasis and satiety. RS found in potatoes can be increased by using certain cooking methods and serving temperatures. The purpose of this trial will compare the acute glycemic and satiety responses after consuming potatoes differing in RS content that are 1) baked then chilled or 2) boiled and consumed hot in overweight females on two separate occasions.

DETAILED DESCRIPTION:
Potatoes are a low-cost, nutrient-dense dietary staple in the U.S. rich in complex carbohydrates, potassium, magnesium, and fiber, but low in fat and sodium. Starch is the main complex carbohydrate found in potatoes that yields glucose to contribute to overall energy needs. Another type of starch found in potatoes is resistant to amylase hydrolysis in the small intestine which is resistant starch (RS). Trials using RS as a functional ingredient (~15-30 g/day) in healthy and overweight adults resulted in improvements in postprandial glucose, insulin sensitivity, satiety hormone response, and subjective satiety. Limited data exists using RS naturally found in commonly consumed foods, such as potatoes. Altering the cooking methods and serving temperatures of potatoes can influence the amount of RS to impact glucose, satiety hormone response, and subjective satiety. Using a cross-sectional, cross-over design, the aim of this study will determine how potatoes 1) baked and chilled or 2) boiled and consumed hot influence postprandial glycemic parameters, satiety hormones (glucagon-like peptide-1, peptide YY, and glucose-dependent insulinotropic polypeptide), subjective satiety, and subsequent energy intake in overweight females.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese (BMI between 28 and 40 kg/m^2)
* Any race or ethnicity

Exclusion Criteria:

* Diabetes or other metabolic disorder, cancer, or cardiovascular disease
* Smoking
* Pregnant or lactating
* More than 5% weight loss or gain over prior 6 months
* Following a special diet
* Sensitivity or aversion to potatoes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Change in postprandial glucose and insulin concentrations | Change in glucose and insulin concentrations collected 15, 30, 60, and 120 minutes following potato intake
  Postprandial glucose and insulin concentrations will be compared between interventions

SECONDARY OUTCOMES:
Change in postprandial glucagon-like peptide- 1 (GLP-1, pg/mL) concentrations | Change in GLP-1 concentrations collected 15, 30, 60, and 120 minutes following potato intake
  Postprandial changes in GLP-1 will be compared between interventions
Change in postprandial peptide YY (PYY, pg/mL) concentrations | Change in PYY concentrations collected 15, 30, 60, and 120 minutes following potato intake
  Postprandial changes in PYY will be compared between interventions
Change in postprandial glucose-dependent insulinotropic peptide (GIP, pg/mL) concentrations | Change in GIP concentrations collected 15, 30, 60, and 120 minutes folllowing potato intake
  Postprandial changes in GIP will be compared between interventions

OTHER OUTCOMES:
Change in postprandial subjective satiety | VAS measured immediately and 120 minutes following potato intake
  Change in postprandial subjective satiety measured by Visual Analogue Scale (VAS) will be compared between interventions
Change in subsequent energy intake | Subsequent energy intake over 48 hours following potato intake
  Change in subsequent energy intake 48 hours following potato intake will be compared between interventions

CONTACTS AND LOCATIONS:
Overall Officials: Mindy Patterson, PhD, RDN, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No